CLINICAL TRIAL: NCT04642950
Title: A Phase II/III Study of Sargramostim in Patients With Coronavirus Disease-2019 (COVID-19)
Brief Title: A Phase II/III Study of Sargramostim
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nobelpharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NPC-26-1
Record Dates: First submitted 2020-11-19; First posted 2020-11-24 (Actual); Results first posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2021-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — sargramostim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NPC-26 (Experimental): Sargramostim (125 μg) will be administered by inhalation twice daily for 5 days, in principle (up to 10 days) as Add-on treatment to the standard treatment.
  Interventions: Drug: Sargramostim
- NP-26 Placebo (Placebo Comparator): Physiological saline will be administered by inhalation twice daily for 5 days, in principle (up to 10 days) as Add-on treatment to the standard treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sargramostim — 250 μg/vial of sargramostim will be dissolved in 4 mL of physiological saline and 125 μg of which will be administered using inhaler twice daily in approximately 10-15 minutes.
  Other Names: Leukine
  Arms: NPC-26
Drug: Placebo — 2 mL of physiological saline will be administered using inhaler twice daily in approximately 10-15 minutes.
  Arms: NP-26 Placebo

SUMMARY:
This is a randomized, placebo-controlled, double-blind, group comparison, multicenter study to evaluate the efficacy and safety of inhalation administration of sargramostim for 5 days, in principle (up to 10 days) as Add-on treatment to the standard treatment in COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

Japanese male or female subjects who have been confirmed to meet all the following criteria.

1. Hospitalized patients under treatment who were severe acute respiratory syndrome coronavirus 2 [SARS-CoV-2] positive by polymerase chain reaction (PCR) test.
2. Patients with clinically diagnosed pneumonia and a percutaneous oxygen saturation [SpO2] of 93% or less on breathing of room air at bed rest.
3. Patients for whom written informed consent has been obtained from those themselves or the legally acceptable representatives.
4. Patients aged 20 years or older and younger than 85 years at the time of obtaining informed consent.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded. Unless otherwise stated, the following criteria refer to those at the time of screening.

1. Patients who have been participating in other intervention studies, such as studies on unapproved pharmacotherapy, within 90 days prior to screening.
2. Patients who have experienced off-label use of approved drugs (including those for COVID-19 treatment other than steroids as standard treatment) within 7 days prior to screening.
3. Patients who are not expected to survive longer than 24 hours after commencement of study drug administration.
4. Patients who are using invasive ventilator or extracorporeal membrane oxygenation (ECMO).
5. Patients who have a chronic respiratory disease requiring continuous home oxygen therapy or ventilator use.
6. Patients with an underlying condition that is considered very unlikely to withdraw ventilator (e.g., motor neuron disease, Duchenne muscular dystrophy, rapidly progressive interstitial pulmonary fibrosis).
7. Patients who have a disease including bronchial asthma, lower respiratory tract infections, and interstitial lung diseases that may affect the assessment of the clinical study, since before the symptom onset of COVID-19.
8. Patients who have a disease including leukemia and leukocytosis that causes leukocytosis.
9. Patients who have a chronic kidney disease requiring dialysis.
10. Patients who have severe liver failure (Child Pugh grade C).
11. Patients aged 80 years or older with any of heart failure, cerebrovascular disease, obesity (BMI 30 or higher), dyslipidemia, hypertension or diabetes.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Japan (7):
  - IUHW Narita Hospital, Narita, Chiba
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama, Kanagawa
  - Japanese Red Cross Society Saitama Red Cross Hospital, Saitama, Saitama
  - St. Luke's International Hospital, Chuo-ku, Tokyo
  - Mishuku Hospital, Meguro-ku, Tokyo
  - Japanese Red Cross Medical Center, Shibuya-ku, Tokyo
  - Center Hospital of the National Center for Global Health and Medicine, Shinjuku-Ku, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shimasaki S, Baba T, Ogura T, Akasaka K, Matsushima H, Izumi S, Takasaki J, Tsushima K, Kinouchi T, Kichikawa Y, Awashima M, Izumo T, Awano N, Nishimura N, Tazawa R, Mikami A, Kitamura N, Ishii H, Kurihara Y, Taniguchi M, Aikawa S, Okada M, Morita Y, Ishikawa Y, Ohinata A, Nakata K. Short-term inhalation of sargramostim with concomitant high-dose steroids does not hasten recovery in moderate COVID-19 pneumonia: a double-blind, randomised, placebo-controlled trial. Infect Dis (Lond). 2023 Dec;55(12):857-873. doi: 10.1080/23744235.2023.2254380. Epub 2023 Oct 6. PMID 37729076

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NPC-26 | NP-26 Placebo
Started | 47 | 23
Completed | 44 | 23
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NP-26 Placebo | NPC-26 | Total
Number analyzed (Participants) | 23 | 47 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 35 | 56
  >=65 years | 2 | 12 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (8.3) | 54.1 (12.5) | 54.7 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 14 | 38 | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Japan | 23 | 47 | 70

OUTCOME MEASURES:

1. Primary Outcome: 2-rank Improvement on a 7-point Ordinal Scale
Description: Number of days to achieve at least 2-rank improvement on a 7-point ordinal scale from baseline until Day 28.
Time Frame: Period until Day 28 (including the case after discharge).
Measure: Median (95% Confidence Interval); unit: Number of Days
Arm/Group | NPC-26 | NP-26 Placebo
Number analyzed (Participants) | 47 | 23
Number of Days | 9 [8 to 9] | 8 [7 to 10]

2. Secondary Outcome: Changes From Baseline in Alveolar-arterial Oxygen Partial Pressure Gradient (A-aDO)
Description: Changes from baseline in alveolar-arterial oxygen partial pressure gradient (A-aDO) on Day 5 and at the end of administration.
Time Frame: Period until Day 28 (including the case after discharge).
Reporting Status: Not Posted

3. Secondary Outcome: Number of Days Until Discharge From Baseline
Description: Number of days until discharge from baseline (days of shifting to Category 7 on a 7-point ordinal scale).
Time Frame: Period until Day 28 (including the case after discharge).
Reporting Status: Not Posted

4. Secondary Outcome: Proportion of Subjects Whose Category Has Shifted to Category 1 or 2
Description: Proportion of subjects whose category has shifted to Category 1 or 2 on a 7-point ordinal scale from baseline until Day 28
Time Frame: Period until Day 28 (including the case after discharge).
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Day1-28
Arm/Group | NPC-26 | NP-26 Placebo
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/23
Serious Adverse Events (participants affected / at risk) | 2/47 | 0/23
Other Adverse Events (participants affected / at risk) | 22/47 | 8/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NPC-26 (N=47) | NP-26 Placebo (N=23)
Myocardial infarction (Cardiac disorders) | 1 | 0 — Acute inferior myocardial infarction
COVID-19 pneumonia (Infections and infestations) | 1 | 0 — Deterioration of COVID-19 pneumonia
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NPC-26 (N=47) | NP-26 Placebo (N=23)
Constipation (Gastrointestinal disorders) | 7 | 4
Hepatocellular injury (Hepatobiliary disorders) | 3 | 0
White blood cell count increased (Investigations) | 7 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 1
Insomnia (Psychiatric disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-04-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT04642950/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/50/NCT04642950/SAP_001.pdf